CLINICAL TRIAL: NCT00579917
Title: Cognitive Behavioral Intervention for BMT/SCT Survivors: Looking Forward
Brief Title: Behavioral Intervention For BMT/SCT Survivors
Acronym: BMT/SCT
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Derald H. Ruttenberg Cancer Center (Unknown); Icahn School of Medicine at Mount Sinai (Other); Hackensack Meridian Health (Other)
Responsible Party: Katherine Duhamel, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-139
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Hodgkin's Disease; Leukemia; Multiple Myeloma; Non-Hodgkin's Lymphoma
Keywords: Survivor; Behavioral Intervention; Bone Marrow; Stem Cell Transplantation
MeSH Terms: conditions — Hodgkin Disease; Leukemia; Multiple Myeloma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1 Cognitive-behavioral therapy (CBT): Cognitive-behavioral therapy (CBT) involves one-on-one counseling
  Interventions: Behavioral: Cognitive Behavioral Therapy: Questionnaires
- 2 Usual Care: Usual Care
  Interventions: Behavioral: Usual Care: Questionnaires

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy: Questionnaires — CBT, we will interview you again after you have completed the 10 sessions. We call these follow-up interviews, and they include several phone calls and a questionnaire you would be asked to complete and then mail in. Each follow-up interview will take between 60 and 210 minutes. If you wish, these follow-up interviews can be done over different days. We will do the follow-up interviews three times; at approximately 4 months, 7 months, and 10 months after you complete the baseline interview.
  Groups: 1 Cognitive-behavioral therapy (CBT)
Behavioral: Usual Care: Questionnaires — If you receive Usual Care, you will not receive CBT while you are in the study. You will complete the questionnaires at the same time as participants who receive CBT. If you receive Usual Care you will be offered 10 sessions of CBT at no charge at the end of the study.
  Groups: 2 Usual Care

SUMMARY:
The purpose of this study is to understand how to help survivors of bone marrow transplant and stem cell transplant (BMT/SCT) with emotional distress. BMT/SCT has become a more common type of treatment for cancer or hematological disorder (blood disease). For this reason, there is concern that adjustment after treatment may be difficult for many persons. We have found that about 25% of BMT/SCT survivors still feel anxious and distressed about their illness and its treatment after at least one year following transplant. This study is one of the first to study the impact of counseling on BMT/SCT survivors. The study is being carried out at Memorial Sloan-Kettering Cancer Center, Mount Sinai Medical Center, and Hackensack University Medical Center.

DETAILED DESCRIPTION:
The use of bone marrow and stem cell transplantation (BMT/SCT) in the treatment of cancer has increased five-fold over the last decade. Among the cancers treated with BMT/SCT are Hodgkin's Lymphoma, non-Hodgkin's Lymphoma, multiple myeloma, and leukemias such as acute lymphoblastic (ALL), acute myelogenous (AML), chronic lymphocytic (CLL), and chronic myelogenous (CML). With the development of non-myeloablative transplants (either "mini" or reduced intensity transplants) for patients unable to tolerate standard BMT/SCT, the use of this procedure is expected to increase substantially over the next five years. BMT/SCT adversely affects almost every aspect of the patient's life (1;2). A standard (fully ablative) transplant involves conditioning with dose intensive chemotherapy, with or without total body irradiation.

Although various medical regimens and supportive psychosocial services are used to reduce the intensity of these side effects, symptoms may persist. Moreover, the drugs used to control side effects often have aversive side effects of their own. Thus, patients must tolerate a protracted course of treatment that is highly aversive and invasive at a time when their lives are disrupted and they are fearful about their survival. A common complaint among survivors is that such problems go unaddressed, and these types of adjustment problems appear to become most intense in the first year post treatment, when physical functioning has stabilized and contact with the BMT/SCT clinical care team wanes (5;10).

ELIGIBILITY:
Inclusion Criteria:

* Have significant psychological distress measured by either:

  * PTSD ONLY - score of 1.0 standard deviation above the mean on the PTSD Checklist-Civilian (PCL-C), or score meets PCL-C symptom cluster criteria for 3 symptom clusters (i.e. re-experiencing, numbing and avoidance combined, and hyperarousal) or 4 symptom clusters (i.e., re-experiencing, numbing only, avoidance only, and hyperarousal); or
  * DISTRESS WITH SOME PTSD - score meets clinically significant impairment on the Brief Symptom Inventory (BSI) global distress index and score meets PCL-C symptom cluster criteria for at least one PCL-C symptom cluster of 3 symptom clusters (i.e. re-experiencing, numbing and avoidance combined, and hyperarousal) or 4 symptom clusters (i.e., re-experiencing, numbing only, avoidance only, and hyperarousal)
* Do not have a substance abuse disorder
* Do not have cognitive impairment as indicated by a score of 3 or lower on the Mini-Mental Status Exam
* Absence of psychotic symptomatology
* Do not have active suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Test the efficacy of a ten-session cognitive-behavioral intervention (CBT-BMT/SCT) on cancer-specific anxiety, psychological distress, and quality of life concerns among BMT/SCT survivors. | conclusion of study

SECONDARY OUTCOMES:
Explore the influence of patient and medical factors on the impact of CBT-BMT/SCT. | conclusion of study

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org